CLINICAL TRIAL: NCT04044768
Title: A Phase 2 Single Arm Open-Label Clinical Trial of ADP-A2M4 SPEAR™ T Cells in Subjects With Advanced Synovial Sarcoma or Myxoid/Round Cell Liposarcoma
Brief Title: Spearhead 1 Study in Subjects With Advanced Synovial Sarcoma or Myxoid/Round Cell Liposarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: USWM CT, LLC (Industry)
Responsible Party: Sponsor
Organization: USWM, LLC (dba US WorldMeds) (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP 0044-002
Record Dates: First submitted 2019-07-09; First posted 2019-08-05 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Synovial Sarcoma; Myxoid Liposarcoma
Keywords: Cell Therapy; T Cell Therapy; SPEAR T Cell; Sarcoma; MRCLS; MAGE A-4; Immuno-oncology
MeSH Terms: conditions — Sarcoma, Synovial; Liposarcoma, Myxoid; Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous genetically modified afamitresgene autoleucel (previously ADP-A2M4) SPEAR™ T cells (Experimental)
  Interventions: Genetic: afamitresgene autoleucel (previously ADP-A2M4)

INTERVENTIONS:
Genetic: afamitresgene autoleucel (previously ADP-A2M4) — Single infusion of autologous genetically modified afamitresgene autoleucel (previously ADP-A2M4) Dose: 1.0 x109 to 10x109 transduced by a single intravenous infusion

SUMMARY:
This is a study to investigate the efficacy and safety of ADP-A2M4 in HLA-A*02 eligible and MAGE-A4 positive subjects with metastatic or inoperable (advanced) Synovial Sarcoma (Cohort 1, 2 and 3 ) or MRCLS (Cohort 1) .

ELIGIBILITY:
Key Inclusion Criteria

* Age ≥16 (10 years at selected sites) and <=75 years
* Diagnosis of advanced synovial sarcoma (Cohort 1, Cohort 2 and Cohort 3) or myxoid liposarcoma / myxoid round cell liposarcoma (Cohort 1 only) confirmed by cytogenetics.
* Previously received either an anthracycline or ifosfamide containing regimen.
* Measurable disease according to RECIST v1.1 prior to lymphodepletion
* HLA-A*02:01, HLA-A*02:02, HLA-A*02:03 or HLA-A*02:06 positive
* Tumor shows MAGE-A4 expression confirmed by central laboratory. North America Only (United States and Canada): Tumor (either an archival specimen or a fresh biopsy) shows MAGE-A4 expression of ≥1+ staining in ≥10% of the cells by immunohistochemistry.
* ECOG Performance Status of 0 or1. For subjects aged ≥10 to ≥16 years old:

Lansky Score ≥60%.

• Left ventricular ejection fraction (LVEF) ≥50%.

Note: other protocol defined Inclusion criteria may apply

Key Exclusion Criteria:

* HLA-A*02:05 in either allele
* Received or plans to receive the following therapy/treatment prior to leukapheresis or lymphodepleting chemotherapy: Cytotoxic chemotherapy, Tyrosine kinase inhibitor (TKI) (e.g. pazopanib), Immune therapy (including monoclonal antibody therapy, checkpoint inhibitors,), Anti-cancer Vaccine, Gene therapy using an integrating vector (subjects who have received a gene therapy using a lentiviral vector may be eligible for the study), Corticosteroids or any other immunosuppressive therapy, Investigational treatment or interventional clinical trial, Allogeneic hematopoietic stem cell transplant, Radiotherapy to the target lesions, Major surgery
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to fludarabine, cyclophosphamide or other agents used in the study.
* History of autoimmune or immune mediated disease
* Symptomatic CNS metastases including leptomeningeal disease.
* Other prior malignancy that is not considered by the Investigator to be in complete remission
* Clinically significant cardiovascular disease
* Uncontrolled intercurrent illness
* Active infection with human immunodeficiency virus, hepatitis B virus, hepatitis C virus, or human T cell leukemia virus
* Pregnant or breastfeeding

Note: other protocol defined Exclusion criteria may apply.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2038-04-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dejka Araujo, MD, Principal Investigator — MD Anderson Cancer Center; Houston TX 77030
Locations (26):
- United States (17):
  - City of Hope, Duarte, California
  - Stanford Cancer Center, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - National Cancer Institute, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Vanderbilt, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutch, Seattle, Washington
  - Medical College of WI Froedtert Hospital, Milwaukee, Wisconsin
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- France (3):
  - Centre Leon Berard, Lyon
  - Hospital Haut Leveque, CHU Bordeaux, Pessac
  - Gustave Roussy Cancer Center, Villejuif
- Spain (3):
  - Hospital Universitari Vall D'Hebron, Barcelona, Catalonia
  - Start Madrid-FJD, Fundación Jimѐnez Díaz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (2):
  - UCLH Cancer Clinical Trials Unit, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Background] D'Angelo SP, Araujo DM, Abdul Razak AR, Agulnik M, Attia S, Blay JY, Carrasco Garcia I, Charlson JA, Choy E, Demetri GD, Druta M, Forcade E, Ganjoo KN, Glod J, Keedy VL, Le Cesne A, Liebner DA, Moreno V, Pollack SM, Schuetze SM, Schwartz GK, Strauss SJ, Tap WD, Thistlethwaite F, Valverde Morales CM, Wagner MJ, Wilky BA, McAlpine C, Hudson L, Navenot JM, Wang T, Bai J, Rafail S, Wang R, Sun A, Fernandes L, Van Winkle E, Elefant E, Lunt C, Norry E, Williams D, Biswas S, Van Tine BA. Afamitresgene autoleucel for advanced synovial sarcoma and myxoid round cell liposarcoma (SPEARHEAD-1): an international, open-label, phase 2 trial. Lancet. 2024 Apr 13;403(10435):1460-1471. doi: 10.1016/S0140-6736(24)00319-2. Epub 2024 Mar 27. PMID 38554725
- [Derived] Sanderson JP, Crowley DJ, Wiedermann GE, Quinn LL, Crossland KL, Tunbridge HM, Cornforth TV, Barnes CS, Ahmed T, Howe K, Saini M, Abbott RJ, Anderson VE, Tavano B, Maroto M, Gerry AB. Preclinical evaluation of an affinity-enhanced MAGE-A4-specific T-cell receptor for adoptive T-cell therapy. Oncoimmunology. 2019 Nov 24;9(1):1682381. doi: 10.1080/2162402X.2019.1682381. eCollection 2020. PMID 32002290

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 2, single-arm, open-label study of afamitresgene autoleucel in HLA-A*02+ participants with MAGE-A4 expressing metastatic or inoperable (advanced) synovial sarcoma or myxoid/round cell liposarcoma (MRCLS) (Cohort 1). Eligible participants received between 1.0 × 10^9 to 10.0 × 10^9 transduced cells of afamitresgene autoleucel, administered as a single IV infusion following lymphodepletion with fludarabine and cyclophosphamide.
Pre-assignment Details: NOTE: Cohort 1 participant Flow, demographics and efficacy cut off was 29Aug2022; Cohort 1 safety cut off was 29Mar2023
Groups:
- Synovial Sarcoma: Eligible participants with metastatic or inoperable (advanced) synovial sarcoma received afamitresgene autoleucel as a single infusion in Cohort 1 (as of data cut off)
- MRCLS: Eligible participants with metastatic or inoperable (advanced) MRCLS received afamitresgene autoleucel as a single infusion in Cohort 1 (as of data cut off)
Period: Overall Study
Arm/Group | Synovial Sarcoma | MRCLS
Started | 44 | 8
Received Afamitresgene Autoleucel | 44 | 8
Completed | 36 (Completed = exited Interventional phase) | 8 (Completed = exited Interventional phase)
Not Completed | 8 | 0
Not completed — Ongoing in Interventional phase at data cut-off | 8 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received T-cell infusion in cohort 1 as of data cut off
Groups:
- Total: Total of all reporting groups
Arm/Group | Synovial Sarcoma | MRCLS | Total
Number analyzed (Participants) | 44 | 8 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 8 | 49
  >=65 years | 3 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (13.07) | 43.4 (12.22) | 41.4 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 2 | 24
  Male | 22 | 6 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 38 | 5 | 43
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 39 | 6 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) (Cohort 1)
Description: Percentage of participants with confirmed tumor response (complete [CR] or partial [PR] response) to treatment as assessed using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by Independent Radiologist review (Cohort 1)
Time Frame: From T-cell infusion until disease progression/recurrence as of data cut off (up to 2 years). Response was assessed at Week 4, Week 8, Week 12, Week 16, and Week 24, and every 2 months +/- 28 days until confirmed disease progression.
Population: Participants who received afamitresgene autoleucel
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Synovial Sarcoma | MRCLS
Number analyzed (Participants) | 44 | 8
percentage of participants | 38.6 [24.36 to 54.50] | 25.0 [3.19 to 65.09]

2. Secondary Outcome: Adverse Events (AE) Including Serious Adverse Events (SAE), SAE, and Adverse Events of Special Interest (AESI) (Cohort 1)
Description: An AE was defined as any untoward medical occurrence in a subject or clinical study participant temporally associated with the use of the study intervention, whether or not considered related to the study intervention. Therefore, an AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. The number of participants with AEs (including SAE), SAE and AESI including cytokine release syndrome, neurotoxicity, ICANS, prolonged cytopenia are presented.
Time Frame: AEs, SAEs, and AESIs were collected at each visit from the start of lymphodepletion of the first subject until the last subject discontinued the interventional phase in cohort 1 as of the safety cut off (up to 3.2 years).
Population: Participants who received afamitresgene autoleucel
Measure: Count of Participants; unit: Participants
Arm/Group | Synovial Sarcoma | MRCLS
Number analyzed (Participants) | 44 | 8
Participants
  AE including SAE | 44 | 8
  SAE | 23 | 3
  AESI - cytokine release syndrome | 33 | 4
  AESI- ICANS | 1 | 0
  AESI- Prolonged cytopenia at Week 4 | 9 | 1

3. Secondary Outcome: The Number of Participants With Replication Competent Lentivirus (RCL)
Description: The presence of RCL was assessed by qPCR targeting a segment of the vesicular stomatitis virus glycoprotein (VSV G) coding sequence.
Time Frame: From T-cell infusion to months 3, 6, and 12 post-infusion, then annually post-infusion (up to 2.8 years as of the data cut off).
Population: Participants who received afamitresgene autoleucel and had a sample tested for VSV-G by qPCR (RCL) at or after 3 months post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Synovial Sarcoma | MRCLS
Number analyzed (Participants) | 31 | 6
Participants | 0 | 0

4. Secondary Outcome: Insertional Oncogenesis (IO)
Description: Deoxyribonucleic acid (DNA) from participants peripheral blood mononuclear cell (PBMC) samples was subjected to lentiviral vector integration site analysis by next-generation sequencing, thus evaluating both the clonality status of the transduced cell population and the genomic localization of individual integration sites. The count of participants with integration sites representing more than 5% of all unique sites is presented.
Time Frame: From 10 months post T-cell infusion up to 20 months post T-cell infusion (as of the data cut off)
Population: Participants who received afamitresgene autoleucel and had a sample analyzed for IO
Measure: Count of Participants; unit: Participants
Arm/Group | Synovial Sarcoma | MRCLS
Number analyzed (Participants) | 9 | 2
Participants | 0 | 0

5. Secondary Outcome: Best Overall Response (BOR) (Cohort 1)
Description: BOR is the best response recorded from the start of T-cell infusion until disease progression/recurrence as assessed by Independent Radiologist review. Response categories are confirmed CR, confirmed PR, stable disease and confirmed progressive disease (PD). Best overall response is a stable disease, if CR or PR are unconfirmed.
Time Frame: From T-cell infusion until disease progression/recurrence as of data cut off (up to 2.6 years). Response was assessed at Week 4, Week 8, Week 12, Week 16, and Week 24, and every 2 months +/- 28 days until confirmed disease progression.
Population: Participants who received afamitresgene autoleucel
Measure: Count of Participants; unit: Participants
Arm/Group | Synovial Sarcoma | MRCLS
Number analyzed (Participants) | 44 | 8
Participants
  Complete Response | 0 | 0
  Partial Response | 17 | 2
  Stable Disease | 23 | 4
  Progressive Disease | 4 | 2

6. Secondary Outcome: Time to Response (TTR) (Cohort 1)
Description: TTR was defined as the interval (weeks) from the date of T-cell infusion to the earliest date of the first documented confirmed CR or confirmed PR as assessed by Independent Radiologist review. TTR (in weeks) = [date of initial confirmed CR or PR - date of T-cell infusion + 1]/7.
Time Frame: From T-cell infusion until first documented confirmed CR or confirmed PR. Response was assessed at Week 4, Week 8, Week 12, Week 16, and Week 24, and every 2 months +/- 28 days until confirmed disease progression.
Population: Participants who received afamitresgene autoleucel and had a confirmed CR or confirmed PR as of data cut off.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Synovial Sarcoma | MRCLS
Number analyzed (Participants) | 17 | 2
Weeks | 4.9 [4.286 to 8.286] | 6.2 [4.286 to 8.143]

7. Secondary Outcome: Duration of Response (DoR) (Cohort 1)
Description: DoR (in months) is defined as ((date of PD (or censoring) - date of initial confirmed CR/PR + 1)/365.25)*12 as assessed by Independent Radiologist review.
  Outcome Measure not yet reached as participants are ongoing in study
Time Frame: From initial confirmed response (CR or PR) until PD (or censored date) as of data cut off.
Reporting Status: Not Posted

8. Secondary Outcome: Progression Free Survival (PFS) (Cohort 1)
Description: PFS is defined as the time from T-cell infusion to the date of the first documentation of PD or death due to any cause, whichever occurs first, as assessed by Independent Radiologist review. PFS (in weeks) was calculated as (date of PD/death [or censored date] - first T-cell infusion date + 1)/7.
Time Frame: From T-cell infusion until first documented PD or death due to any cause (or censored date), whichever occurs first, as of data cut off (up to 2.6 years). Response was assessed at Week 4, 8,12,16, 24, and every 2 months until confirmed PD
Population: Participants who received afamitresgene autoleucel
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Synovial Sarcoma | MRCLS
Number analyzed (Participants) | 44 | 8
Weeks | 16.4 [12.000 to 25.286] | 10.6 [3.714 to 32.000]

9. Secondary Outcome: Overall Survival (OS) (Cohort 1)
Description: OS is defined as the time from the date of T-cell infusion to the date of death (due to any reason) or censored date. OS in months was calculated as ((death date - first T-cell infusion date + 1)/365.25)*12.
  Outcome Measure not yet reached as participants are ongoing in study
Time Frame: From T-cell infusion to death due to any reason (or censored date) as of data cut off (up to 2.6 years).
Reporting Status: Not Posted

10. Secondary Outcome: Peak Persistence (Cohort 1)
Description: Peak persistence of afamitresgene autoleucel cells was reported as vector copy numbers per microgram of genomic DNA from peripheral blood mononuclear cell (PBMC).
Time Frame: From T-cell infusion to 3.2 years (as of data cut off).
Population: Participants who received afamitresgene autoleucel
Measure: Median (Full Range); unit: DNA copies/microgram
Arm/Group | Synovial Sarcoma | MRCLS
Number analyzed (Participants) | 44 | 8
DNA copies/microgram | 229562.050 [18552.9 to 635824.4] | 203534.150 [63586.2 to 346468.3]

11. Secondary Outcome: Time Taken to Achieve Peak Expansion of Genetically Engineered T-cells in PBMCs
Description: Time taken to achieve peak expansion of genetically engineered T-cells in PBMCs by flow cytometry
Time Frame: 2.5 years
Reporting Status: Not Posted

12. Secondary Outcome: Quantitation of Genetically Engineered T-cells in PBMCs
Description: Quantitation of genetically engineered T-cells in PBMCs by flow cytometry
Time Frame: 2.5 years
Reporting Status: Not Posted

13. Secondary Outcome: Time Taken to Achieve Peak Expansion of Genetically Engineered T-cells in PBMCs
Description: Time taken to achieve peak expansion of genetically engineered T-cells in PBMCs by qPCR
Time Frame: 2.5 years
Reporting Status: Not Posted

14. Secondary Outcome: In Vitro Diagnostic (IVD) Assay for Screening
Description: Development and validation of the MAGE-A4 antigen expression companion diagnostic assay
Time Frame: 2.5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected at each visit from the start of lymphodepletion of the first subject until the last subject discontinued the interventional phase in cohort 1 as of the safety cut off (up to 3.2 years).
Description: Adverse events are reported for all participants who received afamitresgene autoleucel
Arm/Group | Synovial Sarcoma | MRCLS
All-Cause Mortality (participants affected / at risk) | 24/44 | 7/8
Serious Adverse Events (participants affected / at risk) | 23/44 | 3/8
Other Adverse Events (participants affected / at risk) | 44/44 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synovial Sarcoma (N=44) | MRCLS (N=8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Empyema (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 4 | 1
Pyrexia (General disorders) | 1 | 1
Influenza-like illness (General disorders) | 1 | 0
Respiratory complication associated with device (General disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Superior vena cava occlusion (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Synovial Sarcoma (N=44) | MRCLS (N=8)
Lymphocyte count decreased (Investigations) | 34 | 6
White blood cell count decreased (Investigations) | 30 | 4
Neutrophil count decreased (Investigations) | 26 | 6
Platelet count decreased (Investigations) | 10 | 2
Alanine aminotransferase increased (Investigations) | 5 | 1
Weight decreased (Investigations) | 5 | 1
C-reactive protein increased (Investigations) | 3 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 4 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 0
Nausea (Gastrointestinal disorders) | 29 | 4
Constipation (Gastrointestinal disorders) | 14 | 5
Vomiting (Gastrointestinal disorders) | 16 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 3
Diarrhoea (Gastrointestinal disorders) | 9 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 0
Fatigue (General disorders) | 15 | 3
Pyrexia (General disorders) | 13 | 1
Non-cardiac chest pain (General disorders) | 10 | 0
Asthenia (General disorders) | 7 | 0
Chills (General disorders) | 7 | 0
Oedema peripheral (General disorders) | 7 | 0
Chest pain (General disorders) | 6 | 0
Pain (General disorders) | 3 | 0
Cytokine release syndrome (Immune system disorders) | 29 | 3
Anaemia (Blood and lymphatic system disorders) | 18 | 4
Lymphopenia (Blood and lymphatic system disorders) | 13 | 1
Neutropenia (Blood and lymphatic system disorders) | 14 | 0
Leukopenia (Blood and lymphatic system disorders) | 9 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 12 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 2
Headache (Nervous system disorders) | 8 | 2
Dizziness (Nervous system disorders) | 5 | 2
Presyncope (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Hypotension (Vascular disorders) | 9 | 0
Hypertension (Vascular disorders) | 7 | 0
Embolism (Vascular disorders) | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Tachycardia (Cardiac disorders) | 6 | 1
Sinus tachycardia (Cardiac disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT04044768/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT04044768/SAP_001.pdf